CLINICAL TRIAL: NCT06282562
Title: FeelFit: High-intensity Interval Training to Improve Self-reported Physical Fitness in Brain Tumor Patients: a Randomized Controlled Trial
Brief Title: FeelFit: High-intensity Interval Training to Improve Self-reported Physical Fitness in Brain Tumor Patients
Acronym: FeelFit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Linda Douw, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL84223.018.23
Record Dates: First submitted 2024-02-06; First posted 2024-02-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Brain Tumor, Primary; Exercise
MeSH Terms: conditions — Brain Neoplasms; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIIT (Experimental): The intervention group will perform High-Intensity Interval Training (HIIT), consisting of two supervised exercise sessions per week on a stationary bike, for 12 weeks.
  In addition, participants will receive information on general guidelines for weekly physical activity levels and will be asked to keep an exercise diary.
  Interventions: Other: High-Intensity Interval Training (HIIT)
- Waiting-list (No Intervention): The control group on the waiting list will be given the option to perform High-Intensity Interval Training (HIIT) after their participation in the study.
  In addition, also participants from the waiting-list control group will receive information on general guidelines for weekly physical activity levels and will be asked to keep an exercise diary.

INTERVENTIONS:
Other: High-Intensity Interval Training (HIIT) — Individualized High-Intensity Interval Training (HIIT) program with two exercise sessions per week for 12 weeks. The exercise sessions will be conducted on a stationary bike, with intensity tailored to each participant's maximum exercise capacity.
  Arms: HIIT

SUMMARY:
The FeelFit study aims to assess the effectiveness of High-Intensity Interval Training (HIIT) in improving self-reported physical fitness in adult brain tumor patients during periods of stable disease, as compared to a waiting-list control group. Furthermore, several secondary and exploratory outcomes will be evaluated. The study is part of the GRIP (GuaRding quality survivorshiP) project, which aims to improve quality of life in brain tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* reduced self-reported physical fitness;
* minimum age of 18 years;
* diagnosed with a primary brain tumor;
* stable disease, i.e. no signs of radiological or clinical tumor progression;
* no oncological treatment for at least two months prior to inclusion;
* able to speak, read and write in Dutch.

Exclusion Criteria:

* Karnofsky Performance Score < 70;
* already participated in a HIIT program < 1 month prior;
* contraindication of exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Self-reported physical fitness | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Self-reported physical fitness is measured using the first question of the International Fitness Scale (IFIS) on general physical fitness, on a 5-point scale where a higher score corresponds to better self-reported physical fitness.

SECONDARY OUTCOMES:
Self-reported fitness | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  In addition to the first question of the International Fitness Scale (IFIS), the other questions about cardiorespiratory fitness, muscle strength, speed and flexibility will also be asked as secondary outcomes.
VO2max | Baseline versus post-intervention (12 weeks)
  Physical fitness defined as the maximal oxygen uptake measured with a cardiopulmonary exercise test.

OTHER OUTCOMES:
Daily physical activity | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  International Physical Activity Questionnaire (IPAQ). A higher score corresponds to a physically more intense activity.
Health-related quality of life questionnaire | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC-QLQ_C30) consists of 30 items and includes five functional scales, three symptom scales, a global health status/quality of life scale, and several single items assessing additional symptoms. The subscales are scored from 0-100 with higher scores representing better quality of life, better functioning, or a higher symptom burden.
Perceived functional impairments | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Work and Social Adjustment Scale (WSAS), consisting of 5 questions on a 8-point scale.
Self-efficacy | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Exercise Self-Efficacy Scale (ESES), consisting of 10 questions on a 4-point scale. A higher score indicates higher exercise self-efficacy.
Mastery | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Pearlin Mastery Scale (PMS), consisting of 7 items on a 4-point scale.
Brain tumor specific quality of life questionnaire | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-BN20, specific for brain tumor patients.
Subjective Happiness | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Subjective Happiness Scale (SHS), consisting of 4 questions on a 7-point scale.
Subjective cognitive functioning | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog), consisting of 37 items on a 5-point scale. A higher score means better cognitive functioning.
Subjective cognitive failure | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Cognitive Failure Questionnaire (CFQ), consisting of 25 items on a 5-point scale. A higher score refers to more cognitive errors.
Fatigue questionnaire | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Checklist Individual Strength (CIS20), consisting of measurements of fatigue severity, concentration problems, reduced motivation, and reduced activity.
Sleep questionnaire | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Pittsburg Sleep Quality Index (PSQI) assesses sleep dysfunction over 1-month interval.
Anxiety questionnaire | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Beck Anxiety Index (BAI), consisting of 21 questions on a 4-point scale.
Self-reported depression questionnaire | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  Beck Depression Index (BDI-PC), consisting of 21 questions on a 4-point scale.
Depression questionnaire | Baseline versus post-intervention (12 weeks) and versus follow-up (12 weeks and 6 weeks follow-up)
  The Center for Epidemiologic Studies Depression questionnaire, consisting of twenty questions regarding symptoms of depression on a 4-point scale.
Muscle strength | Baseline versus post-intervention (12 weeks)
  Hand-held dynamometer
Subjective physical fitness | Baseline versus post-intervention (12 weeks)
  FitMax questionnaire, consisting of thee questions about the maximum capacity of walking, climbing, and cycling, estimating the VO2max.
Objective neurocognitive functioning | Baseline versus post-intervention (12 weeks)
  Neuropsychological assessment (NPA), assessing different brain functions.
Objective neurological functioning | Baseline versus post-intervention (12 weeks)
  Neurological assessment in neuro-oncology scale (NANO). A quantitative evaluation of 9 relevant neurologic domains.
Brain imaging (optional) | Baseline versus post-intervention (12 weeks)
  MRI (magnetic resonance imaging)
Brain activity (optional) | Baseline versus post-intervention (12 weeks)
  MEG (magnetoencephalography)

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Centers, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No